CLINICAL TRIAL: NCT02064426
Title: A Controlled, Parallel Group, Open-label, Multicenter Extension Study to Investigate Efficacy and Safety of Oral BAY85-3934 and Active Comparator (Epoetin Alfa / Beta) in the Long-term Treatment of Subjects With Anemia Associated With Chronic Kidney Disease Who Are on Dialysis in the United States and Japan
Brief Title: Long Term Extension Study for the Maintenance Treatment of Anemia Associated With Chronic Kidney Disease (CKD) in Hemodialysis Subjects on Epoetin Alfa / Beta Treatment Versus BAY85-3934
Acronym: DIALOGUE5
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16209
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Renal Insufficiency, Chronic
Keywords: Anemia of CKD on dialysis
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — molidustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Molidustat (BAY85-3934) (Experimental)
  Interventions: Drug: Molidustat (BAY85-3934)
- Epoetin alfa/beta (Active Comparator)
  Interventions: Biological: Epoetin alfa/beta

INTERVENTIONS:
Drug: Molidustat (BAY85-3934) — Subjects will continue with the same treatment they were receiving in the parent study (16208). BAY85-3934 will be administered daily as oral tablets. Dose assessments will be made every 4 (± 1) weeks. At the scheduled visits, the dose may be titrated on an individualized basis taking into account the subject's Hb response and the tolerability of the previous dose. Total treatment time is up to 36 months. Planned doses include 15, 25, 50, 75, 100, and 150 mg once daily.
  Arms: Molidustat (BAY85-3934)
Biological: Epoetin alfa/beta — Subjects will continue with the same treatment they were receiving in the parent study (16208). Epoetin alfa / beta will be administered as intravenous (IV) or subcutaneous (SC) injections per individual subject regimen according to the local label. Dose assessments will be made every 4 (± 1) weeks. At the scheduled visits,dose may be titrated on an individualized basis taking into account the subject's Hb response and the tolerability of the previous dose.Total treatment time is up to 36 months.
  Arms: Epoetin alfa/beta

SUMMARY:
Evaluate efficacy and safety up to 36 months of titrated dose treatment with BAY85-3934 versus epoetin alfa/beta. Titration will be based on the subject's hemoglobin (Hb) response and tolerability of the prior dose. Planned doses include 15, 25, 50, 75, 100,and 150 mg once daily.

ELIGIBILITY:
Inclusion Criteria:

* Eligible male or female subjects were previously enrolled in Study 16208, have a diagnosis of anemia associated with CKD, and are on hemodialysis.
* Men who agree to use adequate contraception when sexually active or women without childbearing potential
* Participation and completion of treatment in Study 16208; subjects must have received 16 weeks of study medication and completed the end of treatment visit (Day 113) in the parent study
* Mean Hb concentration of 9.5 to 11.5 g/dL, inclusive, during the evaluation period (i.e., the last 4 weeks of the parent study) when the subject completed 16 weeks of treatment with BAY85-3934, epoetin alfa, or epoetin beta in Study 16208

Exclusion Criteria:

* A scheduled kidney transplant or any other organ transplant within the next 6 months (being on a waiting list does not exclude the subject)
* Updates to medical and surgical history which meet the exclusion criteria in the parent study
* Subjects treated with immunosuppressive therapy and the breast cancer resistant protein (BCRP) substrates, irinotecan, topotecan, methotrexate, imatinib, and lapatinib
* Sustained, poorly controlled arterial hypertension or hypotension at baseline, defined as mean BP ≥ 180/110 mmHg or systolic BP < 95 mmHg, respectively
* Severe rhythm or conduction disorder (e.g., HR < 50 or > 110 bpm, atrial fibrillation or flutter, prolonged QT > 500 msec, second or third degree atrioventricular [AV] block)
* New York Heart Association Class III or IV congestive heart failure
* Severe hepatic insufficiency (defined as alanine aminotransferase [ALT], aspartate aminotransferase [AST], or gamma-glutamyl transferase > 3 x the upper limit of norma [ULN], total bilirubin > 2 mg/dL, or Child-Pugh B or C) or active hepatitis in the investigator's opinion
* An ongoing SAE from Study 16208 that is assessed as related to study drug
* Alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2016-10-19 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory hemoglobin level from baseline | Baseline up to 36 months
Number of participants with serious adverse events as a measure of safety and tolerability | Up to 36 months

SECONDARY OUTCOMES:
Maintenance in hemoglobin target range (10.0 to 11.0 g/dL) | Up to 36 months
Maintenance in hemoglobin target range (9.5 to 11.5 g/dL) | Up to 36 months
Duration of treatment exposure | Up to 36 months
Number of subjects requiring titration of dose | Up to 36 months
Change of reticulocyte count from baseline of this study | Baseline up to 36 months
Change of reticulocyte count from baseline of study 16208 | Baseline up to 36 months
Change of red blood cell count from baseline of this study | Baseline up to 36 months
Change of red blood cell count from baseline of study 16208 | Baseline up to 36 months
Change of hematocrit from baseline of this study | Baseline up to 36 months
Change of hematocrit from baseline of study 16208 | Baseline up to 36 months
Change of central laboratory hemoglobin level from baseline of this study | Baseline up to 36 months
Change of central laboratory hemoglobin level from baseline of study 16208 | Baseline up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- United States (19):
  - Azusa, California
  - Long Beach, California
  - Lynwood, California
  - Northridge, California
  - San Dimas, California
  - Whittier, California
  - New Port Richey, Florida
  - Pembroke Pines, Florida
  - Detroit, Michigan
  - Creve Coeur, Missouri
  - Buffalo, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Grand Prairie, Texas
  - Houston, Texas
  - Mansfield, Texas
- Japan (3):
  - Muroran, Hokkaido
  - Kuwana, Mie-ken
  - Kyoto

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/